CLINICAL TRIAL: NCT07083934
Title: Comparison of Ultrasound Guided Supraclavicular Brachial Plexus Block With and Without Peripheral Nerve Stimulation (PNS) Guidance: A Randomized Controlled Tria
Brief Title: Ultrasound-Guided Supraclavicular Block With vs Without PNS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-9043-30909
Record Dates: First submitted 2025-06-13; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Supraclavicular Plexus Block; Ultrasound; Anaesthesia

STUDY DESIGN:
Intervention Model Description: 2 groups assignment
  1. Ultrasound and nerve stimulator
  2. Only Ultrasound
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (US) (Active Comparator): Use of an ultrasound guidance device without a peripheral nerve stimulator for nerve block placement. Only ultrasound will be used for the procedure.
  Interventions: Device: No peripheral nerve stimulator
- Ultrasound+PNS (Experimental): Use of a peripheral nerve stimulator device in combination with ultrasound for nerve block placement.
  Interventions: Device: Peripheral nerve stimulator

INTERVENTIONS:
Device: Peripheral nerve stimulator — Peripheral nerve stimulator along with ultrasound
  Arms: Ultrasound+PNS
Device: No peripheral nerve stimulator — No peripheral nerve stimulator with ultrasound. Only ultrasound will be used
  Arms: Ultrasound (US)

SUMMARY:
Peripheral Nerve Blockade (PNB) became reliable with the advent of Ultrasound (US) and Peripheral Nerve Stimulation (PNS).

US offers real-time visualization but has limitations, especially with deep or obscured nerves.

PNS complements US by confirming nerve proximity through motor responses. Combining both may enhance safety and success of nerve blocks. This study compares US-guided blocks with and without PNS in a randomized trial.

DETAILED DESCRIPTION:
Peripheral Nerves Blockade (PNB) via local anaesthetics is a method of providing anesthesia and analgesia to the limbs and it was well established in the late 20th century. However, it did not come very well into practice because of unreliability, high rate of complications and failure due to lacking of accurate and reliable techniques of nerve localization at that point in time. It was only when newer nerve localization methods, such as Peripheral Nerve Stimulation (PNS) and Ultrasound (U/S) Imaging started becoming commercially available that the trend of Regional Anaesthesia started getting recognized among the physicians. PNB as a sole anaesthesia technique for limb surgery took further integration in practice and widespread acceptance among anaesthetist in the last decade, once ultrasound technology advanced to newer heights resulting in compact and more mobile units, higher resolution, needle recognition software etc.

When compared to PNS guided regional anaesthesia (PGRA), ultrasound guided regional anaesthesia (UGRA) offers a number of important practical advantages such as direct real-time visualization of the anatomy of interest, needle pathway and its passing through structures and spread of local anaesthetic, and the potential for instantaneous needle re-adjustments as per need. All this allows for safer and more effective distribution of local anaesthetic in the region of desired peripheral nerve. This superiority of Ultrasound Guidance led to fade in the use of PNS guidance in the Regional Anaesthesia practice over the recent years.

Regardless of the previously discussed superiority of U/S Guidance in Regional anaesthesia (RA), it has its own limitations. Such limitations include difficulty in visualization and identifying neural structures when they are lying far away from the skin either due to thick overlying subcutaneous adipose tissue in the obese patients or simply because of the presence of nerve bundle in the deeper tissue planes, and inability to confidently identify and exclude the placement of needle tip within the nerve, where if an injectate is injected will lead to nerve damage.

Such limitations of U/S Guidance in RA can be circumvented by using PNS Guidance in its conjunction. PNS works by delivering a small pulse of electric current through the needle tip which when in close proximity to a neural structure will lead to its stimulation and its respective muscle contraction, thereby helping us in identifying the neural structure of interest. Current density (with pulse duration at 1ms and frequency 2Hz) of around 1 mA for superficial nerves and 1.5-2mA for deeper nerves is enough to elicit a desired motor response. Eliciting a motor response at an even higher current density can be discomforting to the patient as well as misleading to the operator as neural structures can get stimulated through tissues and fascial planes. Similarly, Current density can also be used to predict the intra-fascicular or intraneural needle placement. One study showed that minimum stimulation (Median [interquartile range]) threshold outside was 0.60 mA [0.40-1.0] and inside 0.30 mA [0.20-0.40], where, the difference of 0.30 mA was statistically significant. Therefore, a lower limit for the current density can be used as a safety margin beyond which no muscle activity should be elicited by using PNS.

So, considering the additional benefits of PNS Guidance that it can potentially concur in facilitating UGRA in achieving effective and safer PNB, we propose and design a randomized control trial by comparing the UGRA with and without PNS Guidance in achieving PNB and its outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* ASA physical status I to IV
* No contraindications to regional anaesthesia
* Operative site located at the mid to lower arm, including the elbow, forearm, wrist, or hand
* Ability to provide informed consent
* Ability to reliably report symptoms to the research team related to regional anaesthesia

Exclusion Criteria:

* Patient's refusal to participate.
* Inability to provide first-party consent due to cognitive impairment.
* Cognitive dysfunction which can lead to difficulties in communication and cooperation of patient.
* Preexisting neuropathy.
* Preexisting coagulopathy.
* Patients who will be shifted to ICU due to post - operative ventilatory support.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of peripheral nerve block (PNB) with ultrasound-guided regional anesthesia (UGRA) with and without peripheral nerve stimulation (PNS) | From administration of peripheral nerve block (PNB) until confirmation of successful block onset, assessed up to 60 minutes post-procedure
  Comparison of PNB success rate between UGRA alone and UGRA combined with PNS guidance.

CONTACTS AND LOCATIONS:
Overall Officials: Azhar Rehman, Mbbs Fcps, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
It will be shared among investigatots only

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT07083934/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT07083934/ICF_001.pdf